



## Consent Form.

Study title: Understanding the nature of the safety and quality of care problems experienced by service users accessing community-based mental health services: a qualitative study.

Once you have read the participant information sheet and asked the researcher about any questions you have, please write your initials in each box and sign your name to show you agree with the items below:

| No. | Item | Initials |
|---|---|---|
| 1. | I confirm that I have understood the Participant Information Sheet (dated: [DATE AND | |
| | <b>VERSION NUMBER]</b> ) for this study. I have had the opportunity to ask questions and these | |
| | were answered satisfactorily. | |
| 2. | I understand that I may not be able to take part in the study if I do not give consent to any | |
| | one element on this form. | |
| 3. | I understand that taking part in this study is voluntary, and that I am able to withdraw at | |
| | any time before or during the interview or focus group. | |
| 4. | I understand that I can withdraw the data from my interview for up to two weeks after | |
| | taking part in the study, up until a cut-off date of [TWO WEEKS AFTER DATE OF | |
| | SCHEDULED INTERVIEW]. I understand that if I take part in a focus group, it will not be | |
| | possible to withdraw my data after I have taken part, due to the nature of the group | |
| | discussion. | |
| 5. | I agree that direct quotes from my interview or focus group can be used in written | |
| | reporting of this research. I understand that my personal details will not be used and that | |
| | it will not be possible to identify me from any publications of the study findings. | |
| 6. | I consent to my interview or focus group being audio-recorded and transcribed by an | |
| | external company (outside of the University), who will do this task whilst maintaining | |
| | confidentiality. | |
| 7. | I understand that if I tell the research team anything which suggests: a risk of harm to | |
| | myself or others, unreported staff malpractice, or unreported incidents of criminal | |
| | activity, that they will need to share this information with the relevant agency. I am aware | |
| | that the research team will discuss this with me first. | |
| 8. | I have had enough time to decide to participate. | |
| 9. | I agree to take part in this study. | |







The following items are about whether or not you would like to be contacted about the results of this study, or to be informed about future opportunities to get involved with research conducted by this team. There items are optional, and if left blank we will assume you do not agree.

| No. | Item | Initials |
|---|---|---|
| 10. | I would like to be informed about the results of this study. | |
| 11. | I would like to be updated about the wider research project being conducted by this | |
| | research team entitled 'Improving safety and quality of mental healthcare', including | |
| | being notified about future opportunities to shape research, or to take part in a study. | |

| Name of participant | Date | Signature |
|-------------------------------|------|-----------|
| | / / | |
| Name of person taking consent | Date | Signature |
| | / / | |

**Chief Investigator:** Dr Claire Henderson; **Lead Researcher:** Phoebe Averill, <u>phoebe.averill@kcl.ac.uk</u>.

1 copy to the participant, 1 copy to the research team.